CLINICAL TRIAL: NCT02910895
Title: Development of a Platform of Patient Derived Xenografts (PDX) and 2D/3D Cell Cultures of Soft Tissue Sarcomas (STS): Protocol to Obtain Tumour Material From Patients With STS.
Brief Title: A Platform of Patient Derived Xenografts (PDX) and 2D/3D Cell Cultures of Soft Tissue Sarcomas (STS)
Acronym: SarcomaPDX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N16STS; NL58626.031.16 (Registry Identifier: CCMO)
Record Dates: First submitted 2016-07-21; First posted 2016-09-22 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Sarcoma; Xenograft Model; 2D/3D Cell Cultures
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): single tumor biopsy
  Interventions: Other: tumor biopsy

INTERVENTIONS:
Other: tumor biopsy — biopsy

SUMMARY:
Outside the setting of well-designed prospective clinical studies, the current standard preoperative RT should be a conventionally 1.8-2 Gy fractionated regimen to a total dose of 50 Gy in 5-6 weeks. However, given the vast diversity of sarcoma subtypes, it is also unlikely to assume a uniform therapeutic management to be optimal for all sarcomas alike. Other than 2 Gy fraction sizes and/or 50 Gy total dose series have been investigated in the past and should be further exploited in the future, but the practical implementation in humans is hampered by the rarity of the disease.

The current systemic treatment of sarcomas consists of both the older cytotoxic chemotherapies and the newer targeted therapies like tyrosine kinase inhibitors. But it is hard to predict which patients will respond to which specific systemic treatment. This leads to worse prognoses and unnecessary toxicity for sarcoma patients. Despite the fact that the number of sarcoma patients in current studies is too small with a mix of different subtypes, some subtypes show a better response than other subtypes. This platform may form the basis for preclinical translational investigations with radiotherapy and various systemic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosed (non-) metastatic intermediate to high grade STS
* Local recurrences are allowed
* Age ≥ 18 years
* Able and willing to undergo tumour biopsies or tumour sampling during surgery
* Localization of sarcoma enables safe biopsy or surgery
* Written informed consent

Exclusion Criteria:

* Known coagulation disorder and/or anticoagulant medication in as far it might interfere with a safe biopsy procedure (to the discretion of the treating physician and attending radiologist)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
A platform of Patient Derived Xenografts (PDX) of Soft Tissue Sarcomas of patients with sarcomas | 4 months
  take rate
The take-rate of fresh human PDX tumour material in nude mice. | 4 months
  take rate
A consistent system for further anti-sarcoma therapy (both RT and chemotherapy experiments) | 2 years after start of study
  take rate
A platform of 2D/3D cell cultures (organoids) of Soft Tissue Sarcomas. | 6 weeks
  take rate
A model for translational research | 2 years after start of study
  take rate

SECONDARY OUTCOMES:
The passage possibilities of human PDX tumour material by freezing, storing, thawing and re-inoculating in nude mice | 4 months after implantation of tumour material
  take rate of continuous growth of implantation of tumor material
Fractionation sensitivity on several STS subtypes in PDX. | 4 months
  take rate
To study the passage possibilities of 2D/3D cell cultures by freezing, storing and thawing | 1 month
  take rate of continuous growth

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No